CLINICAL TRIAL: NCT05218135
Title: Evaluation of the Current Care Processes for Stroke Care in Flemish Hospitals Via a Breakthrough Improvement Collaborative
Brief Title: BIC: Evaluation of the Current Care Processes for Stroke Care in Flemish Hospitals
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kris Vanhaecht, Professor, KU Leuven
Other Study IDs: BIC4Stroke
Record Dates: First submitted 2022-01-18; First posted 2022-02-01 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Breakthrough improvement collaborative
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Learning session 1: explain key interventions, explain BIC methodology, retrospective patient record analysis Learning session 2: feedback report, share best practices, discussion, set priorities, teaching and improvement, retrospective patient record analysis Learning session 3: feedback report, share best practices, discussion, set priorities, teaching and improvement, retrospective patient record analysis Learning session 4: feedback report

SUMMARY:
Different studies showed large variation between care processes in multiple diseases, which lead to large variation in outcomes. Better adherence to evidence-based guidelines for these diseases can reduce this variation and can improve the health outcomes. Since international studies have demonstrated wide variations in care processes for acute stroke, it would be interesting to repeat these investigations in the population of stroke patients. Worldwide, stroke is a leading cause of disability and death. Every two seconds, someone across the world experiences a symptomatic stroke. 50% of stroke survivors has moderate to severe neurologic deficits, 25% of them depend on others. In Belgium, stroke is one of the most important causes of invalidity. Every year approximately 18 000 people in Belgium experiences a stroke, which results in almost one person every two hours, with a mortality rate of 30%. The world health organization has the ambition to significantly reduce the mortality and risk factors for non-communicable diseases by 2025. The mortality and disability in stroke patients can be reduced by organized stroke care, which includes effective strategies in stroke management, treatment and prevention. Also, other health domains, like functional recovery, healthcare costs and patient satisfaction, were positively related to adherence on stroke guidelines. This evidence had been converted in several clinical guidelines for stroke care. However, the adherence to these guidelines is variable. As already mentioned before, international studies have demonstrated wide variations in care processes for acute stroke. However, a positive relationship has been shown between the implementation of evidence-based clinical guidelines and the quality of stroke care. Therefore, it is important to both implement these guidelines and to improve the adherence to them.

The aim of this study is to map the variation in stroke care in Flemish hospitals and to get an overview about the variation within and between these hospitals. During this study, electronic patient records will be analyzed to check which interventions are performed in a specific patient and of which no information could be found in de patient record.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Admitted to the emergency department and diagnosed with an ischemic stroke

Exclusion Criteria:

* Diagnosed with cerebral venous thrombosis
* Diagnosed with hemorrhage
* Thrombectomy performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 2610 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Variation within and between hospitals | through study completion, an average of 3 months
  Variation of Brain imaging + timing, Glycemia (venous blood sample or finger prick) + timing, Clinical neurologic examination + timing, Time of onset, Administration of IV tPA + timing, Administration of aspirin + timing Blood pressure, time of first measurement and measurement frequency during first 72h, Oxygen saturation, time of first measurement and measurement frequency during first 72h, Temperature, time of first measurement and measurement frequency during first 72h, Glycemia and measurement frequency during first 72h, First dysphagia screening and timing, Advice from speech therapist if screening failed and timing, Cardiac monitoring, Screening for depression, ADL screening, The use of a bladder catheter is not recommended, Prophylactic treatment with antibiotics is not recommended, Deep venous thrombosis prevention

SECONDARY OUTCOMES:
Mortality rate | Through study completion on average of 3 months
  Mortality rate
modified Rankin Scale | Through study completion on average of 3 months
  modified Rankin Scale going from 0 (no symptoms) until 6 (death)

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No